CLINICAL TRIAL: NCT00139802
Title: Low Restenosis Rate of the NIR Coronary Stent: Results of the Danish Multicenter Stent Study (DANSTENT) - a Randomized Study Comparing a First-Generation With a Second-Generation Stent.
Brief Title: DANish Multicenter STENT Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DANSTENT
Record Dates: First submitted 2005-08-30; First posted 2005-08-31 (Estimated); Last update posted 2005-08-31 (Estimated); Status verified 1997-01

CONDITIONS: Ischemic Heart Disease; Stable Angina; Unstable Angina
MeSH Terms: conditions — Myocardial Ischemia; Angina, Stable; Angina, Unstable

INTERVENTIONS:
Device: Coronary Stent Implantation

SUMMARY:
The purpose of the study was to evaluate procedural and late outcome of coronary artery stenting using 2 different unmounted stents

ELIGIBILITY:
Inclusion Criteria:

* Stable, unstable or silent angina,
* De novo lesion

Exclusion Criteria:

* Allergy to ticlopidine
* Recent myocardial infarction
* Expected survival > 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400
Dates: Start 1997-04; Study Completion 2001-06

CONTACTS AND LOCATIONS:
Overall Officials: Henning Kelbaek, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Copenhagen, Denmark

REFERENCES:
- [Result] Jorgensen E, Kelbaek H, Helqvist S, Jensen GV, Saunamaki K, Kastrup J, Madsen JK, Klovgaard L, Thuesen L, Villadsen A, van Weert AW, Reiber JH; Danish multicenter stent study (DANSTENT). Low restenosis rate of the NIR coronary stent: results of the Danish multicenter stent study (DANSTENT)--a randomized trial comparing a first-generation stent with a second-generation stent. Am Heart J. 2003 Feb;145(2):e5. doi: 10.1067/mhj.2003.32. PMID 12595860